CLINICAL TRIAL: NCT04765761
Title: Efficacy of Proseal Laryngeal Mask Airway With or Without Introducer-tool Stabilization for Pressure Controlled Ventilation in Adults Undergoing Elective Surgery: a Randomized Controlled Study
Brief Title: Proseal Laryngeal Mask Airway With or Without Introducer-tool Stabilization for Pressure Controlled Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Ganga Ram Hospital (Other)
Responsible Party: Principal Investigator, Nitin Sethi, DNB, Senior Consultant, Sir Ganga Ram Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EC/01/21/1800
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Airway Remodeling
MeSH Terms: conditions — Airway Remodeling

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated into 2-groups. Group-1 will be the 'PLMA with Introducer' group and group-2 will be the 'PLMA without Introducer' group.
Who Masked: Participant
Masking Description: The patient will be blinded to the study intervention as designated by the randomized group he/she would be allocated to. The investigator however will not be blinded to the group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLMA with Introducer' (Active Comparator): PLMA placed in position with the help of the introducer-tool and then the introducer-tool retained in place throughout the institution and duration of positive pressure ventilation.
  Interventions: Device: PLMA with introducer
- PLMA without Introducer (Active Comparator): PLMA placed in position with the help of the introducer-tool and then the introducer-tool removed before institution of positive pressure ventilation.
  Interventions: Device: PLMA without introducer

INTERVENTIONS:
Device: PLMA with introducer — The pro-seal laryngeal mask airway (PLMA) will be inserted along with introducer tool which will be kept in-situ throughout the duration of positive pressure ventilation
  Arms: PLMA with Introducer'
Device: PLMA without introducer — The pro-seal laryngeal mask airway (PLMA) will be inserted along with introducer tool which will be removed after insertion and patient will be ventilated using PLMA without the introducer in-situ throughout the duration of positive pressure ventilation
  Arms: PLMA without Introducer

SUMMARY:
ProSeal laryngeal mask airway (PLMA) has become an effective alternative to tracheal tube for gaining airway access and for the institution and maintenance of positive pressure ventilation (PPV) in patients undergoing short-to-moderate duration (20-60 minutes) surgery under GA. The PLMA is the more preferred supra-glottic airway access device for advantages therein over the other SGA's, including having an option of dedicated introducer-tool (ease of placement), availability of esophageal opening (allows regurgitated fluid to bypass the airway), and reinforced main body tube (prevents luminal compression). Additionally, as compared to other supra-glottic airway devices, the PLMA device has been found to be more consistent in providing PPV to patients' lungs during GA. However, not uncommonly, PLMA itself is not consistent in maintaining trouble-free PPV owing to the vulnerability to position change, especially secondary to the rhythmic movement posited by back pressure during PPV. This movement vulnerability induced by PPV may be because of the size/shape of PLMA cuff that does fit upon placement but gets vulnerable to undue movement during PPV.

We hypothesize that keeping the introducer-tool in position after insertion of PLMA result in greater stabilization of PLMA in position by minimizing the movement that occurs due to back-pressure effect on the cuff during positive pressure ventilation. This randomized study intends to evaluate whether keeping the introducer-tool in position (after PLMA insertion) accords greater positional stabilization to the PLMA and thereby offers greater efficacy for achieving adequate pressure control ventilation in paralyzed anesthetized adults undergoing elective surgery.

DETAILED DESCRIPTION:
Supraglottic airways (SGA) have become a standard proposition in management of the upper airway. These devices have suitably interposed its utility as airway conduit between the facemask and the tracheal tube in terms of anatomical position and degree of invasiveness. These devices sit outside of trachea but provide a hands-free means of achieving a gas-tight airway. In the year 1989, the first SGA, the classic laryngeal mask airway (C-LMA), became available. As time went on, additional variants of LMA came into use.

The ProSeal Laryngeal mask airway (PLMA), introduced in 2000, is by far the most specialized SGA device. It comprises of four main subparts: the cuff, inflation line with pilot balloon, airway tube, and the gastric drain tube. All components are made of silicone and are latex-free. Studies indicate that size 3/4 is most preferable for adult women and size 4/5 for adult men.

The airway (breathing, ventilation) tube of the PLMA is shorter and smaller in diameter than its C-LMA counterpart. PLMA's wire-reinforced body makes it more flexible and yet resistant to luminal compression. The locating-strap on the anterior distal tube of PLMA prevents finger slipping off the tube and also provides an insertion slot for an 'introducer-tool'. An additional safety accessory vent under the drainage tube in the bowl help avoid secretions from pooling and accessing the upper airway. The PLMA has a deeper bowl than C-LMA and has a bite-block between the airway and drain tubes at the level of teeth to prevent device injury.

In a correctly positioned PLMA, the cuff tip lies behind the cricoid cartilage at the origin of the esophagus; allows liquids/gases a bypass escape from the stomach and reduces the risk of gastric insufflation, regurgitation and pulmonary aspiration; and provides information about the PLMA position. The drain tube is designed to prevent the epiglottis from occluding the airway tube, thus eliminating the need for aperture bars. A gastric tube, doppler probe, temperature probe can be passed into the oesophagus through the drainage port.

The PLMA also has a second dorsal cuff which pushes the mask anteriorly to provide a better seal around the glottic aperture.

As per the standard guidelines, an introducer-tool (a curved, malleable, silicone-coated blade with a guiding handle) is used to facilitate placing an PLMA in the pharyngo-laryngeal slot, and helps greatly with the first-insertion placement success.

Once in place, the PLMA offers a dependable conduit through which effective PPV can be instituted. Interestingly, although the PLMA placement and position adequacy has a static corollary to it and that the institution of PPV situates a dynamic airflow system; not uncommonly, there are problems to effective PPV even through an adequately placed PLMA. The rhythmic PPV which leads to back pressure onto the PLMA cuff often result in subtle cuff movements resulting in leak at the desired PPV pressure.

Based on past clinical data in unit regarding safety of this procedure we hypothesize that keeping the introducer-tool in position (after facilitating insertion of PLMA) minimizes unwanted position changes owing to back pressure effect of PPV on the PLMA cuff, and therefore, would enable us to achieve and maintain adequate ventilation during GA.

We plan this study with an objective to compare efficacy of PLMA with or without introducer tool assisted stabilization during PPV in anaesthetized paralyzed patients undergoing short to moderate duration surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20 - 60 years.
2. ASA physical status I and II.

Exclusion Criteria:

1. Patients having complaints of acid-peptic disease, chronic constipation, feeling of stomach fullness after meal.
2. Previous gastrointestinal surgery
3. History of hiatus hernia
4. Known case of substance abuse or chronic alcoholism
5. Psychiatric illness
6. Pregnant patients
7. Anatomical defects of the mandible.
8. Dental problems (Missing teeth, loose teeth)
9. Surgery requiring Trendelenburg position.
10. Surgery requiring position change during procedure
11. Morbid obesity with OSAS.
12. Failure to obtain consent

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal Seal pressure of the PLMA | From time of insertion of PLMA till 120-minutes intraoperatively
  Oropharyngeal seal pressure (in cmH2O) will be measured by closing the expiratory valve of the anaesthetic circle system at a fixed gas flow rate of 3L/min, and noting the equilibrated upper airway pressure

SECONDARY OUTCOMES:
Efficiency of positive pressure ventilation (PPV) | From time of insertion of PLMA till 120-minutes intraoperatively
  It will be determined by calculating the tidal volume generated on institution of PPV and pressures (cmH2O) required to achieve 10ml /kg tidal volume through PLMA.
Postoperative sore throat | From end of surgery till 24 hours postoperatively
  The presence of sore throat will be graded on a two-point scale; 0: sore throat absent, 1: sore throat present
Postoperative cough | From end of surgery till 24 hours postoperatively
  The presence of cough will be graded on a two-point scale; 0: cough absent, 1: cough present
Postoperative difficulty in swallowing | From end of surgery till 24 hours postoperatively
  The presence of difficulty in swallowing will be graded on a two-point scale; 0: difficulty in swallowing absent, 1: difficulty in swallowing present
Postoperative difficulty in speaking | From end of surgery till 24 hours postoperatively
  The presence of difficulty in speaking will be graded on a two-point scale; 0: difficulty in speaking absent, 1: difficulty in speaking present
Quantitative assessment of positive pressure ventilation (PPV) | From time of insertion of PLMA till 120-minutes intraoperatively
  The positive pressure ventilation will be adjudicated as "trouble-free PPV" if there is no leak and the tidal ventilation is achieved (as reflected by consistent EtCO2 tracings) with standardized ventilation parameters (f- 14, I:E- 1:2, Inspiratory pressure- 20cm H20).
  The positive pressure ventilation will be adjudicated as "trouble-prone PPV" if there is a leak around PLMA and the tidal ventilation could not be achieved with standardized ventilation parameters (frequency- 14, I:E- 1:2, Inspiratory pressure- 20cm H20) but can finally be achieved with routine adjustments.
  The positive pressure ventilation will be adjudicated as ''failed positive pressure ventilation'' wherein it is not possible to establish PPV through the PLMA conduit despite maximum adjustments

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Saxena, MBBS, MD, Study Chair — Sir Ganga Ram Hospital, New Delhi, INDIA; Amitabh Dutta, MD, PGDHR, Principal Investigator — Sir Ganga Ram Hospital, New Delhi, INDIA; Abishek SS, Principal Investigator — Sir Ganga Ram Hospital, New Delhi, INDIA; Manish Kohli, DA, DNB, Principal Investigator — Sir Ganga Ram Hospital, New Delhi, INDIA
Locations (1):
- Nitin Sethi, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No